CLINICAL TRIAL: NCT05635747
Title: A 90 Day Observational Study as an Extension to the Phase 3, Open Labeled, Exploratory Study of RELiZORB to Evaluate Safety, Tolerability, and Nutrient Absorption in Children With Short Bowel Syndrome Who Are Dependent on PN
Brief Title: A 90 Day Observational Study as an Extension to the Phase 3,Open Labeled Exploratory Study of RELiZORB
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Alcresta Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Puder, MD, PhD, Professor Pediatric General Surgery, Boston Children's Hospital
Other Study IDs: P00042824
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Short Bowel Syndrome; Malabsorption
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients who have completed the Relizorb Trial and consented into the 90 day extension trial: Patients aged 2-18 who have completed the 90 day open label phase 3 Relizorb trial who consent to the 90 day observational Relizorb extension trial
  Interventions: Device: Relizorb Enzyme Cartridge

INTERVENTIONS:
Device: Relizorb Enzyme Cartridge — Tube feeds run across device to digest fats.

SUMMARY:
Children with inadequate intestinal absorption due to loss of large amounts of small bowel require intravenous nutrition (feeding through the vein) to sustain hydration and nutrition to avoid starvation and dehydration; however, intravenous (IV) nutrition can lead to complications including liver failure. Tube feeding directly to the small intestine avoids the complications of IV nutrition, but fats are not fully digestible due to inadequate bowel function. We propose to predigest the fat using a small cartridge attached to the feeding tube to allow for rapid absorption with the possibility of reducing or eliminating the need for intravenous nutrition. Goal of the observational study is to determine safety and tolerability of Relizorb Enzyme Cartridge for an additional 90 days after the original trial

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is often due to the loss of large amounts of small intestine that compromises digestive absorption. The treatments include (1) a high-calorie diet that includes vitamins, minerals, carbohydrates, proteins and fats; (2) injections of vitamins and minerals; (3) administration of drugs to slow the normal movement of the intestine or to increase the surface area of the intestinal lining; and (4) feeding through the vein (i.e., parenteral nutrition or PN). Many patients cannot wean from PN due to reduced intestinal length or function. Patients on long-term PN frequently experience serious metabolic complications, sepsis, hepatic biliary disorders including cholestasis, and fibrosis and can progress to liver failure. Full intestinal feeding (enteral nutrition) without PN is the optimal way to prevent the above complications.

Enterally administered long chain triglycerides in patients with SBS, especially those with hepatic dysfunction, are not well tolerated due to bile acid malabsorption, which leads to decreased micelle formation and fat digestion. The dietary fat is unable to be emulsified by the bile acids and acted on by lipases before exiting the patient as stool. Switching to other forms of fat such as medium-chain triglycerides (MCTs) that do not require micelles for absorption may be better tolerated in patients with bile acid or pancreatic insufficiency but are not optimal as they increase the osmotic load in the intestine. This may increase the chance of stool dumping; moreover, MCTs do not contain essential fatty acids (FAs). The ability to provide the essential FAs such as those present in enteral formulas in a form that does not require the formation of micelles for absorption, would allow patients with SBS and those who are no longer PN dependent to receive adequate nutrition and continue to maintain the same growth trajectory as when they received the majority of their nutrition parenterally.

RELiZORB is a digestive enzyme cartridge connected in-line with enteral feed tubing sets designed to mimic the function of pancreatic lipase. It is hypothesized that by using an external lipase device (RELiZORB) enteral nutrition will be better absorbed, and PN dependence reduced as enteral autonomy is increased. This product uniquely eliminates the need for intestinal emulsification and lipase activity and eliminates the risk of drugs, including lipases, allowing absorption at the time the diet enters the gut. The device has been shown to digest >90% of fat in most enteral formulas.

Goal of the observational study is to determine safety and tolerability of Relizorb Enzyme Cartridge for an additional 90 days after the original trial. Patients with short bowel syndrome aged 2-18 who are dependent on parenteral nutrition and enteral feeds who completed the original Relizorb Trial. Participants will continue to use the Relizorb device with enteral nutrition for 90 additional days.

Primary objective:

•To evaluate the effect of the RELiZORB enzyme cartridge when used with enteral nutrition daily for an additional 90 days (for a total of 180 days from enrollment) on the change from baseline in PN calories.

Secondary objective:

•To evaluate the effect of the RELiZORB enzyme cartridge when used with enteral nutrition daily for an additional 90 days (for a total of 180 days from enrollment) on the change from baseline in body weight

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently enrolled in the ongoing RELiZORB study titled "A 90 day, Phase 3, Open Labeled Exploratory Study of RELiZORB to Evaluate Safety, Tolerability, and Nutrient Absorption in Children with Short Bowel Syndrome who are Dependent on Parenteral Nutrition"
2. The parent or legal guardian of the patient is able to read, understand, and is willing to provide informed consent (and assent, if applicable).
3. The patient (if assent is applicable) or parent or legal guardian of the patient is able to understand the requirements of the study and is willing to bring the patient to all clinic visits and complete all study-related procedures (as determined by the investigator).
4. A parent or legal guardian is willing to provide written authorization for the use and disclosure of protected health information.

Exclusion Criteria:

1. Active clinically-significant pancreatic or biliary disease, as determined by the investigator.
2. Change in patient formula such that the new formula is not compatible with the RELiZORB cartridge (example, insoluble fiber-containing formulas)
3. Determined by the investigator to be unsuitable for participation for any reason.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 32 pediatric subjects with SBS, aged 2 years - 18 years who are PN dependent are expected to be enrolled in the ongoing clinical study and will be invited to participate in this extension study. Eligibility will be established by the investigator based on the inclusion and exclusion criteria for the extension study.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of the RELiZORB enzyme cartridge when used with enteral nutrition daily for an additional 90 days | 90 days
  change from baseline in PN calories

SECONDARY OUTCOMES:
To evaluate the effect of the RELiZORB enzyme cartridge when used with enteral nutrition daily for an additional 90 days | 90 days
  the change from baseline in body weight (weight-for-age z-score).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Puder, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Freedman S, Orenstein D, Black P, Brown P, McCoy K, Stevens J, Grujic D, Clayton R. Increased Fat Absorption From Enteral Formula Through an In-line Digestive Cartridge in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):97-101. doi: 10.1097/MPG.0000000000001617. PMID 28471913